CLINICAL TRIAL: NCT03987503
Title: The No One Waits Study: Acceptability and Feasibility of Community-based Point-of-diagnosis HCV Treatment Study
Acronym: NOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-342-5516
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis C, Chronic
Keywords: People who inject drugs; Homeless; Community-based testing and treatment
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — sofosbuvir-velpatasvir drug combination; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- at Point-of-Diagnosis HCV treatment (Experimental): At the point of HCV infection diagnosis, (HCV RNA positive and anti-HCV positive) individuals who meet eligibility criteria and elect to start HCV treatment at the same visit and monitored at two-week intervals at the community-site.
  Interventions: Drug: Epclusa (SOF/VEL); Device: Fibroscan® 430 Mini Plus
- Passive observation (Active Comparator): Participants who test positive for HCV chronic infection (HCV RNA positive, and anti-HCV positive) but elect to not enroll in the intervention arm. Electronic medical record data will be reviewed for up to 2 years for HCV related care information (e.g., HCV treatment start date, end date, SVR-12).
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Epclusa (SOF/VEL) — a trained physician will provide research participants with two-week supply of SOF/VEL. Treatment is: 1 tablet SOF/VEL (400 mg sofosbuvir/100 mg velpatasvir) daily x 12 weeks. The initial 2-week supply is provided by Gilead Sciences and will be dispensed to participants upon enrollment. Prescriptions and insurance prior authorizations for SOF/VEL will be submitted by the study pharmacist though the UCSF Specialty Pharmacy. The study team will be notified once insurance-authorized drug is available and will bring participants' medication in 2 supplies to the study site prior to study visits.
  Arms: at Point-of-Diagnosis HCV treatment
Drug: Standard of care — Standard of HCV care provided by medical care provider
  Arms: Passive observation
Device: Fibroscan® 430 Mini Plus — Trained research staff will measure participants liver stiffness using liver ultrasonographic elastography. Research staff place ultrasound gel directly on participant's skin on the area of the torso. Research staff will position the participant's body on the exam table to assure the liver can be located, placing the small probe on the body's surface (skin with gel) and begin recording images of the participant's liver.
  The procedure will take 15-30 minutes, depending on the ease with which the research staff is able to accurately locate the participant's liver.
  Results from the FibroScan will be discussed with a trained provider.
  Other Names: Fibroscan
  Arms: at Point-of-Diagnosis HCV treatment

SUMMARY:
Direct-acting antiviral (DAA) therapy for hepatitis C virus (HCV) offers a cure to those with chronic HCV infection. For marginalized communities, linkage to care services often aren't enough to overcome barriers to accessing the medical system. For difficult to link populations, offering treatment at the same non-clinical community space may improve uptake and reduce loss-to-follow-up. The purpose of this 2 year study is to assess the feasibility, acceptability and effectiveness of accelerated initiation of commercially available DAA therapy targeting socially marginalized communities (e.g., medically underserved, homeless, people actively injecting drugs). The study will be carried out at two community sites that perform HCV testing: (a) fixed community site and (b) community mobile site via clinical research van. Participants (n=150) who test anti-HCV positive and HCV RNA positive (chronic infection) are invited to enroll into the no one waits (NOW) Study and begin HCV treatment at point of diagnosis. All evaluation, medication dissemination, and follow-up care will take place at the project site. The investigators will estimate the effect of on-site point-of-diagnosis (POD) treatment on (1) time from HCV testing to treatment initiation, (2) completing treatment, and (3) attaining (sustained virologic response) SVR-12; overall and by study site. A secondary product will be a lesson learned guide of recommendations for implementing a POD on-site test and treat program for dissemination beyond San Francisco.

DETAILED DESCRIPTION:
This study is a non-randomized interventional study.

NOW is an open-label study evaluating the feasibility, acceptability, and effectiveness of an accelerated community-based treatment program of SOF/VEL x 12 weeks started at time of chronic HCV diagnosis (intervention).

The purpose of the proposed study is to assess the feasibility, acceptability and effectiveness of accelerated initiation of commercially available direct-acting antiviral (DAA) therapy targeting socially marginalized communities (e.g., medically underserved, homeless, people actively injecting drugs). The proposed study will be carried out at two community sites that perform HCV testing: (a) fixed community site and (b) community mobile site. The fixed site is located in the Tenderloin Neighborhood of San Francisco: The Quaker Meeting House (QMH). The QMH is the current location for an established drop-in center for young adult (< 30 years old) people who inject drugs, a group at highest risk for acquiring new HCV infection but representing a group with the lowest engagement in HCV treatment. The QMH site is complete with two phlebotomy stations, centrifuge, clinical exam station, interview rooms, and office space. The QMH research site will prioritize study enrollment for young adult people who inject drugs (PWID). The community mobile site (DeLIVER Van) is situated in a mobile van; a 145 sqft space equipped with a phlebotomy station, clinical exam table, centrifuge, and portable Fibroscan® 430 Mini Plus. The DeLIVER Van will serve two neighborhoods in San Francisco with high HCV burden but few community-based medical service organizations: the Bayview neighborhood and Outer Mission neighborhood.

The investigators will (1) implement new tools, notably FIBROSCANS, to measure fibrosis in an at-risk group (HCV positive patients); (2) implement a new standard of care, treatment on-demand in an at-risk group (HCV positive active drug users); (3) assess the feasibility and acceptability of expanding standard of care into non-clinical settings.

At study entry, participants will undergo a combined eligibility screening/entry visit, which includes HCV testing (antibody and RNA), rapid anti-HIV test, and HBsAG (hepatitis B virus surface antigen) testing and consent for medical record linkage. If HCV RNA reactive, participants are offered enrollment into the treatment cohort and provided 2 week supply of SOF/VEL (provided by Gilead as part of the NOW Study) upon completion of a clinical evaluation, baseline survey, and venipuncture for baseline labs. If the participant is actively insured, the study investigators will obtain insurance-authorized SOF/VEL to complete the remainder of the 12 week treatment course. If the participant is not actively insured, the study team will assist with insurance acquisition and subsequently obtain insurance-authorized SOF/VEL to complete the remainder of the 12 week treatment course. For any participants, if insurance-authorized SOF/VEL is delayed beyond the initial 2 week study-provided SOF/VEL, additional supplies of SOF/VEL as needed to ensure an uninterrupted 12 week treatment course. Participants will return every 2 weeks during treatment (12 week course) for medication dispensation and study visit activities. And for two post-treatment visits for clinical monitoring (e.g., HCV RNA testing) and research activities.

Study participants in the intervention study (cohort): Chronic HCV (anti-HCV positive and HCV RNA positive) men and women ages ≥18 years newly diagnosed or re-engaged in care at a fixed or mobile community-based site. Participants should be HBsAg negative, have no known history of decompensated cirrhosis or end stage renal disease, not be pregnant or breastfeeding, and not be taking medications that are contraindicated with SOF/VEL.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* anti-HCV and HCV RNA positive,
* Lifetime injection drug use or blood transfusion before 1991
* interested in starting HCV treatment at the time of diagnosis
* Women of childbearing potential engaged in sexual activity that could lead to pregnancy
* must consent to use contraception and agree to pregnancy testing during treatment
* If currently not enrolled in insurance, agree to assistance to enroll in insurance

Exclusion Criteria:

* HBsAg positive from pre-screening visit and no medically controlled hepatitis B virus (HBV) condition
* History of hepatic decompensation (ascites, hepatic encephalopathy, or variceal hemorrhage).
* Current use of medications that is not compatible with SOF/VEL use, according to current prescribing guidelines, including amiodarone or a proton pump inhibitor exceeding 20 mg of omeprazole equivalent.
* Prior treatment with an NS5a based HCV treatment regimen with subsequent viral rebound. Participants who have clear HCV reinfection as defined by an HCV GT that is different from the original genotype may enroll. If genotype results are not available from the initial and subsequent HCV infection, the individual will not be enrolled unless participant can provide SVR-12 record confirming HCV cure.
* Pregnancy or breastfeeding.
* Life expectancy of < 12 months as assessed by study clinical health provider.
* Late exclusion criteria: Participants with the following lab values at week 0 will be evaluated on a case by case basis for continuation of SOF/VEL at the week 2 visit
* Albumin < 3.0
* Hemoglobin < 8.0 (women) and < 9.0 g/dl ( men)
* Platelet count < 50,000
* creatinine (Cr) clearance (estimated by Cockcroft-Gault) < 30 ml/min
* aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) > 10 x ULN
* Total bilirubin > 1.5x ULN (for participants on atazanavir, > 3 x ULN), international normalized ratio (INR) > 1. 5 x ULN

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan D Morris, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Summary statistics of primary and secondary outcome data and overall sample demographics (e.g., gender, age, ethnicity/race) will be shared with researchers through annual conference presentations and final results related to the study aims will be disseminated via peer-reviewed manuscripts.

REFERENCES:
- [Derived] Kim RG, McDonell C, McKinney J, Catalli L, Price JC, Morris MD. Staff-Facilitated Telemedicine Care Delivery for Treatment of Hepatitis C Infection among People Who Inject Drugs. Healthcare (Basel). 2024 Mar 25;12(7):715. doi: 10.3390/healthcare12070715. PMID 38610138
- [Derived] Morris MD, McDonell C, Luetkemeyer AF, Thawley R, McKinney J, Price JC. Community-Based Point-of-Diagnosis Hepatitis C Treatment for Marginalized Populations: A Nonrandomized Controlled Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2338792. doi: 10.1001/jamanetworkopen.2023.38792. PMID 37862013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 1 2020 and October 31, 2021 street-outreach recruitment targeted people experiencing homelessness and injecting drugs. Eligibility included being 18 years or older and reporting either lifetime injection drug use or having a blood transfusion in or before 1992.
Pre-assignment Details: Of the 492 screened for hepatitis C infection, 403 were excluded. Reasons for exclusion included: 3 untreated HIV, 246 anti-HCV negative, 102 anti-HCV positive and RNA negative, 18 unsuccessful blood draw, 12 other clinical criteria (treatment experience, untreated HIV, HBsAg positivity, or decompensated cirrhosis), and 22 did not return for RNA results. Of the 89 participants eligible for treatment, 87 accepted and 2 declined treatment. All 87 received "at Point-of-Diagnosis HCV Treatment".
Period: Overall Study
Arm/Group | at Point-of-Diagnosis HCV Treatment
Started | 87
Treatment Completion | 69 (Completed 12 weeks of SOF/VEL treatment)
Attended Sustained Virologic Response at 12-weeks (SVR12) Blood Draw Visit | 65
Undetectable Result at SVR12 | 58
Completed | 65 (Achieved sustained virologic response 12 weeks post-treatment (SVR12))
Not Completed | 22
Not completed — Lost to Follow-up | 20
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | at Point-of-Diagnosis HCV Treatment
Number analyzed (Participants) | 87
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [37 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 49
  More than one race | 9
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response at 12-weeks (SVR-12)
Description: The number and percent attaining SVR12 after POD HCV treatment, overall, using an intention to treat (participants taking one or more doses of SOF/VEL) and per-protocol analysis (participants completing treatment).
  Test Details: Blood serum was collected by venipuncture to quantitatively test for HCV RNA. The lower limit of quantification for this polymerase chain reaction test was 15 IU/mL (1.18 log IU/mL) and the minimum level of blood plasma needed was 1.8 mL.
Time Frame: 12 weeks from treatment completion
Population: Participants who started HCV treatment at the point of diagnosis (Intention-to-treat analysis)
Measure: Count of Participants; unit: Participants
Groups:
- Per-Protocol Analysis: Among those who completed 12-week course of treatment
Arm/Group | at Point-of-Diagnosis HCV Treatment | Per-Protocol Analysis
Number analyzed (Participants) | 87 | 69
Participants | 58 | 58

2. Secondary Outcome: Time From Anti-HCV Testing to Treatment Initiation
Description: Time from HCV testing visit to treatment initiation
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- HCV Treatment at the Point of Diagnosis: Participants received HCV treatment at the point of positive RNA and antibody HCV tests.
Arm/Group | HCV Treatment at the Point of Diagnosis
Number analyzed (Participants) | 87
days | 7 [6 to 14]

3. Secondary Outcome: Treatment Completion
Description: Percent of those who started treatment who completed course of treatment
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HCV Treatment at the Point of Diagnosis
Number analyzed (Participants) | 87
Participants | 69

4. Secondary Outcome: Undetectable RNA at Treatment Completion
Description: Percent of people who had undetectable RNA at end of treatment.
  Test Details: Blood serum was collected by venipuncture to quantitatively test for HCV RNA. The lower limit of quantification for this polymerase chain reaction test was 15 IU/mL (1.18 log IU/mL) and the minimum level of blood plasma needed was 1.8 mL.
Time Frame: 12 weeks
Population: Three of the 69 participants could not receive end-of-treatment HCV RNA testing because of blood draw challenges. This is represented in the 61/66 reported with undetectable RNA at treatment completion.
Measure: Count of Participants; unit: Participants
Arm/Group | HCV Treatment at the Point of Diagnosis
Number analyzed (Participants) | 66
Participants | 61

5. Secondary Outcome: Acceptability: Number of Persons Who Decline POD Treatment
Description: Number of persons who decline POD treatment
Time Frame: 1 day
Population: The number of participants analyzed for this endpoint is greater than in other analyses . since were are studying acceptability of the intervention. Specifically, of participants eligible for treatment (n=89), 87 accepted and enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | HCV Treatment at the Point of Diagnosis
Number analyzed (Participants) | 89
Participants | 87

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | HCV Treatment at the Point of Diagnosis
All-Cause Mortality (participants affected / at risk) | 0/87
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT03987503/Prot_SAP_000.pdf